CLINICAL TRIAL: NCT00301873
Title: Phase II Study of Zometa (Zoledronic Acid) to Prevent Osteoporosis in Patients With Brain Tumors
Brief Title: Zoledronate in Preventing Osteoporosis in Patients With Primary Malignant Glioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Novartis (Industry); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00010125; P50NS020023 (NIH)
Record Dates: First submitted 2006-03-09; First posted 2006-03-13 (Estimated); Results first posted 2013-01-16 (Estimated); Last update posted 2013-02-18 (Estimated); Status verified 2013-02

CONDITIONS: Brain Tumors; Osteoporosis; Central Nervous System(CNS)Malignancies
Keywords: osteoporosis; adult anaplastic astrocytoma; adult giant cell glioblastoma; adult anaplastic oligodendroglioma; adult gliosarcoma; adult mixed glioma; recurrent adult brain tumor; adult glioblastoma
MeSH Terms: conditions — Brain Neoplasms; Osteoporosis; Astrocytoma; Glioblastoma; Oligodendroglioma; Gliosarcoma; Glioma | interventions — Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IV Zometa (Experimental): Zometa will be given at 4 mg intravenously over 15 minutes every 3 months for 1 year.
  Interventions: Drug: IV Zometa

INTERVENTIONS:
Drug: IV Zometa — Zometa will be given at 4 mg intravenously over 15 minutes every 3 months for 1 year.
  Other Names: zolondronic acid

SUMMARY:
RATIONALE: Zoledronate may prevent bone loss in patients with primary malignant glioma.

PURPOSE: This phase II trial is studying how well zoledronate works in preventing osteoporosis in patients with primary malignant glioma.

DETAILED DESCRIPTION:
This is an open-labeled trial to determine the incidence of osteoporosis in brain tumor patients and effect of Zometa every three months. Zometa will be given at 4 mg intravenously over 15 minutes every 3 months for 1 year. The patients will undergo a baseline bone densitometry test that will be repeated at six months and one year. Information on the patient's tolerability of Zometa as well as any skeletal-related complications that happen will be collected. Data with respect to the dose and duration of glucocorticoids and anticonvulsants will be collected since both of these therapies have shown to directly affect bone density. Serial markers (N-telopeptide) of bone turn over will be collected at baseline and every 3 months prior to the infusion of Zometa. Karnofsky performance status will be monitored as a function of mobility.

Accrual Goal 60 patients over a 18-month period, averaging 3-4 new enrollees per month. Thirty-five patients to reach the 6-month assessment.

OBJECTIVES:

* To determine the bone mineral density of the patients at baseline and any changes over 12 months while receiving Zometa every 3 months.
* To determine the incidence of skeletal-related complications in this cohort of brain tumor patients.
* To determine the safety and tolerability of Zometa in brain tumor patients.
* To determine the effects of glucocorticoids and anticonvulsants on bone density.

Response Criteria The primary efficacy endpoint will be the patient's bone densitometry, and how it changes over the course of one year of Zometa therapy. The bone densitometry after 6 months and 12 months of Zometa will be compared to the baseline. The secondary efficacy variable will be the prevention of skeletal-related events (compression fracture, any fracture requiring surgery) which given the heterogeneity of the patient population will be a qualitative variable. Date with respect to the dose and duration of glucocorticoids and anticonvulsants will be collected since both of these therapies have shown to directly affect bone density. Serial markers (N-telopeptide) of bone turn over will be collected.

Outcome assessment The patient's bone densitometry will be determined by Dexa-scan at the baseline, after six months of Zometa and after one year of Zometa. The bone density (Dexa- scan) will be reviewed by the outside radiologist or Duke radiology in conjunction with the primary investigator. A decrease of > -0.5 on the T-score will be coded as a treatment failure and patients will be discontinued from the study and referred to Endocrinology or Orthopedic Surgery for best clinical management. In addition, any skeletal-related event (fractures) will be coded as a treatment failure. The patient population will be heterogeneous in terms of their functional capacity, exercise capacity, anticonvulsant and glucocorticoid dos

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically confirmed diagnosis of a primary brain tumor.
2. Patients must be on Depakote ( Valproic Acid) or one of the following enzyme inducing anticonvulsants (EIAC) therapies. Phenobarbital, Dilantin, Trileptal, Tegretol and/or on more than physiologic replacement steroid therapy (Dexamethasone >0.75 mg/d, prednisone >5 mg/d or hydrocortisone >20 mg/d).
3. Age > 18 years.
4. Karnofsky performance score > 60%
5. Adequate renal and liver function as demonstrated by laboratory values performed within 14 days, inclusive, prior to the administration of Zometa, except for the creatinine, which will be within 72 hs of Zometa administration:

   * Serum creatinine < 2.0 mg/dl and calculated creatinine clearance of >60 mL/min
   * Total serum bilirubin < 1.5 times upper limit of laboratory normal
   * Serum glutamoc-oxaloacetic transaminase (SGOT) and serum glutamic pyruvic transaminase (SGPT) < 2.5 times upper limit of laboratory normal
   * Alkaline phosphatase of <2 times upper limit of laboratory normal
6. Patients must have recovered from any effects of major surgery.
7. Patients must have a life expectancy of greater than 12 weeks.
8. Patients or legal guardian must give written, informed consent.

Exclusion Criteria:

1. Patients who are poor medical risks because of non-malignant systemic disease as well as those with acute infection treated with intravenous antibiotics.
2. Previous or concurrent malignancies at other sites with the exception of surgically cured carcinoma in-situ of the cervix and basal or squamous cell carcinoma of the skin.
3. Known HIV positivity or AIDS-related illness.
4. Pregnant or nursing women.
5. Women of childbearing potential who are not using an effective method of contraception. Women of childbearing potential must have a negative serum pregnancy test 72hours prior to administration of study and be practicing medically approved contraceptive precautions.
6. Men who are not advised to use and effective method of contraception.
7. Patients previously diagnosed with osteoporosis requiring oral bisphosphonates.
8. Known hypersensitivity to Zometa® (zoledronic acid) or other bisphosphonates
9. Current active dental problems including infection of the teeth or jawbone osteonecrosis of the jaw (ONJ), of exposed bone in the mouth, or of slow healing after dental procedures.
10. Recent (within 6 weeks) or planned dental or jaw surgery (e.g.. extraction, implants).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-05; Primary Completion 2011-02 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James J. Vredenburgh, MD, Study Chair — Duke University
Locations (1):
- Duke Comprehensive Cancer Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were accrued between February 2006 and January 2008 within the clinic at Duke Comprehensive Cancer Center.
Period: Overall Study
Arm/Group | IV Zometa
Started | 59
Completed | 59
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | IV Zometa
Number analyzed (Participants) | 59
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 49
  >=65 years | 10
Age Continuous [Mean (Standard Deviation); unit: years] | 54.7 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 38
Anticonvulsant use [Number; unit: participants]
  yes | 54
  no | 5
Steroid use [Number; unit: participants]
  yes | 41
  no | 18

OUTCOME MEASURES:

1. Primary Outcome: Percent of Patients With Change in Combined Bone Mass Density T-score <= -0.5.
Description: Percent of patients who failed treatment as defined by a decrease of 0.5 or more from baseline in the combined T-score as measured by Dexa-scan. The patient's bone densitometry was determined by Dexa-scan at baseline, after 6 months of Zometa and after 1 year of Zometa. The t-score, which is a comparison of a person's bone density with that of a healthy 30-year-old of the same sex, was generated by Dexa-scan for the spine and femur. The combined T-score is the minimum of the T-score for the spine and femur. A lower t-score implies a lower BMD.
Time Frame: 6 and 12 months
Population: 59 patients were accrued; however only 27 had a follow-up assessment at 6 months and 19 at 12 months.
Measure: Number; unit: percentage of patients
Arm/Group | IV Zometa
Number analyzed (Participants) | 59
percentage of patients
  At 6 months (n=27) | 3.7
  At 12 months (n=19) | 10.5

2. Secondary Outcome: Skeletal-related Complications
Description: Number of patients who experience skeletal-related complications during the administration of Zoledronate.
Time Frame: 1 year
Population: All patients.
Measure: Number; unit: participants
Arm/Group | IV Zometa
Number analyzed (Participants) | 59
participants | 0

3. Secondary Outcome: Mean Change in Bone Mass Density (BMD)
Description: Mean change in the combined t-score was measured by Dexa-scan. The patients bone density was determined by Dexa-scan at baseline, after 6 months Zometa and after 12 months of Zometa. The t-score, which is a comparison of a person's bone density with that of a healthy 30-year old of the same sex, was generated by Dexa-scan for the spine and femur. A lower t-score implies a lower BMD. The combined t-score is the minimum of the t-score for the spine and that for the femur. BMD change from baseline at 6 and 12 months in the combined t-score was defined as the follow-up combined t-score minus the baseline combined t-score.
Time Frame: 6 & 12 months
Population: 59 patients were accrued to the study; however follow-up at 6 months was available from 27 patients and at 12 months data was available from 19 patients.
Measure: Mean (Standard Deviation); unit: T score units
Arm/Group | IV Zometa
Number analyzed (Participants) | 59
T score units
  Change in combined BMD at 6 months (n=27) | .01 (.21)
  Change in combined BMD at 12 months (n=19) | -.06 (.31)
Statistical Analysis 1: Comparison: IV Zometa; 59 patients were accrued to the study. The 27 patients with follow-up at 6 months are included in an analysis to assess the association between baseline steroid use and bone mass density at 6 months using linear regression; Test type: Superiority or Other; p = .2212, Regression, Linear — The p-value is a test of whether the slope of the regression line is non-zero; The linear regression assesses the relationship between baseline baseline steroid use and BMD change at 6 months (outcome); Slope = -.107, Standard Error of Mean .0855
Statistical Analysis 2: Comparison: IV Zometa; 59 patients were accrued to the study. The 27 patients with follow-up at 6 months are included in an analysis to assess the association between baseline anticonvulsant use and bone mass density at 6 months using linear regression; Test type: Superiority or Other; p = .0413, Regression, Linear — this p-value is at test of whether the slope of the regression line is non-zero; The linear regression assesses the relationship between anticonvulsant use and BMD change at 6 months (outcome); Slope = .2357, Standard Error of Mean .1091
Statistical Analysis 3: Comparison: IV Zometa; 59 patients were accrued to the study. The 19 patients with follow-up at 12 months are included in an analysis to assess the association between baseline steroid use and bone mass density at 12 months using linear regression; Test type: Superiority or Other; p = .0418, Regression, Linear — this p-value is at test of whether the slope of the regression line is non-zero; The linear regression assesses the relationship between baseline steroid use and BMD change at 12 months (outcome); Slope = -.232, Standard Error of Mean .1029
Statistical Analysis 4: Comparison: IV Zometa; 59 patients were accrued to the study. The 19 patients with follow-up at 12 months are included in an analysis to assess the association between baseline anti-convulsant use and bone mass density at 12 months using linear regression; Test type: Superiority or Other; p = .1026, Regression, Linear — the p-value is a test of whether the slope ofl the regression line is non-zero; The linear regression assesses the relationship between anticonvulsant use and BMD change at 12 months; Slope = .2123, Standard Error of Mean .1209

ADVERSE EVENTS:
Time Frame: All Adverse Events regardless of grade over a period of 1 year
Description: Common Terminology for Adverse Events (CTCAE)3.0 used for collecting adverse events (AEs). Converted to 4.0 for this report. Serious Adverse Events(SAE): of the 16 pts affected by an SAE only, 3 were possibly, probably, or definitely related to Zometa. AEs: Of the 27 pts affected by an AE 12 were possibly, probably, or definitely related to Zometa.
Arm/Group | IV Zometa
Serious Adverse Events (participants affected / at risk) | 16/59
Other Adverse Events (participants affected / at risk) | 31/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IV Zometa (N=59)
fever (General disorders) | 5
Skin ulceration (Skin and subcutaneous tissue disorders) | 1
dehydration (Metabolism and nutrition disorders) | 1
diarrhea (Gastrointestinal disorders) | 2
Intracranial hemorrhage (Nervous system disorders) | 1
infections and infestations-other (Infections and infestations) | 3
Skin infection (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 1
Device related infection (Infections and infestations) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 1
Facial nerve disorder (Nervous system disorders) | 1
seizure (Nervous system disorders) | 4
Depressed level of consciousness (Nervous system disorders) | 3
headache (Nervous system disorders) | 3
phlebitis (Vascular disorders) | 1
thrombo embolic event (Vascular disorders) | 3
Vascular access complication (Injury, poisoning and procedural complications) | 2
Neutrophil count decreased (Investigations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IV Zometa (N=59)
fatigue (General disorders) | 14
fever (General disorders) | 3
insomnia (Psychiatric disorders) | 7
rash maculo-papular (Skin and subcutaneous tissue disorders) | 3
anorexia (Metabolism and nutrition disorders) | 4
constipation (Gastrointestinal disorders) | 8
diarrhea (Gastrointestinal disorders) | 5
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 7
ataxia (Nervous system disorders) | 5
cognitive disturbance (Nervous system disorders) | 6
confusion (Psychiatric disorders) | 10
dizziness (Nervous system disorders) | 5
memory impairment (Nervous system disorders) | 11
mood alteration (Psychiatric disorders) | 3
Peripheral motor neuropathy (Nervous system disorders) | 8
Peripheral sensory neuropathy (Nervous system disorders) | 4
seizure (Nervous system disorders) | 3
Depressed level of consciousness (Nervous system disorders) | 5
dysphasia (Nervous system disorders) | 8
blurred vision (Eye disorders) | 3
headache (Nervous system disorders) | 9
arthralgia (Musculoskeletal and connective tissue disorders) | 5
urinary incontinence (Renal and urinary disorders) | 4
erectile dysfunction (Renal and urinary disorders) | 7

LIMITATIONS AND CAVEATS:
Limitations include early pt termination leading to small numbers of subjects analyzed (eg no BMD study at 6 and/or 12 mos)secondary to the poor overall survival (eg median survival 3-9 mos)associated with recurrent glioblastoma multiforme(GBM) pts.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No